CLINICAL TRIAL: NCT04513015
Title: Markers of Oxidative Stress in Inflammatory Bowel Disease in Children and Adults: Risk Factors and Implications for a Dietetic Approach
Brief Title: Markers of Oxidative Stress in Inflammatory Bowel Diseases: Risk Factors and Implications for a Dietetic Approach
Acronym: OxIBDiet
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università Politecnica delle Marche (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Principal Investigator, Carlo Catassi, M.D., Professor, Università Politecnica delle Marche
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OxIBDiet-2020
Record Dates: First submitted 2020-07-27; First posted 2020-08-14 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Inflammatory Bowel Diseases
Keywords: oxidative stress imbalance; antioxidant diet
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: IBD subjects (40 children and 40 adults, 50% with CD and 50% with UC) will be enrolled in different conditions: at diagnosis, in remission, at relapse. For each IBD subject an age and gender matched control subject will be enrolled (40 children and 40 adults).
  In a subgroup of subjects (20 children and 20 adults, 50% with CD and 50% with UC) in clinical remission/mild disease a dietetic approach will be proposed. Patients on steroids and patients with strictures will not be enrolled for this part of the study. Patients will be randomized in 2 groups: Group Antioxidant diet will receive 8 weeks of antioxidant dietary treatment and group Normal diet will continue a normal dietetic scheme (corresponding to a isocaloric, normolipidic diet for age and sex).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antioxidant diet (Experimental): Group Antioxidant diet will receive 8 weeks of antioxidant dietary treatment
  Interventions: Dietary Supplement: Antioxidant diet
- Normal diet (Active Comparator): Group Normal diet will continue a normal dietetic scheme (corresponding to a isocaloric, normolipidic diet for age and sex).
  Interventions: Dietary Supplement: Normal dietetic scheme

INTERVENTIONS:
Dietary Supplement: Antioxidant diet — The "antioxidant diet" will include the principal antioxidant molecules/nutrients previously shown to be beneficial in IBD: Flavonoids, particularly resveratrol and curcumin; Olive oil; Glutathione, Vitamins A, C, E; Carotenoids; Selenium and Omega 3 Fatty Acids (PUFAs). The daily amount of these substances will be calculated following the published evidence, whether these amounts will not be achievable by a standard diet, a supplementary formulation will be proposed.
  Arms: Antioxidant diet
Dietary Supplement: Normal dietetic scheme — Isocaloric, normolipidic diet for age and sex
  Arms: Normal diet

SUMMARY:
Inflammatory bowel disease (IBD), including Crohn's disease (CD), Ulcerative Colitis (UC) and IBD-unclassified (IBD-U) is a chronic inflammatory intestinal disorders that affect both children and adults. Patients with IBD can present with severe gastrointestinal symptoms, require frequent hospitalizations, expensive medical treatments and can develop invalidating complications requiring surgery. The incidence of IBD is increasing worldwide. The pathogenesis is multifactorial with immunological, environmental and genetic factors contributing to the disease. There is evidence that oxidative stress (OS) imbalance is involved in IBD onset and evolution, although the exact contribution to the pathogenes is unclear. An antioxidant dietetic approach is promising as an adjunctive treatment of IBD. The main aims of this project are to characterize the OS imbalance in IBD in relation to disease's features and to genetic factors and to evaluate the efficacy of an antioxidant dietetic treatment

DETAILED DESCRIPTION:
IBD is a complex disorder that is thought to be the result of an aberrant immune response to commensal bacteria in a genetically susceptible host. The chronic inflammation along the gastrointestinal tract that characterizes IBD results from an imbalance of effector lymphocytes and pro-inflammatory cytokines. Some of the cytokines, as well as the triggered leukocytes and activated macrophages, can produce large amounts of reactive oxygen species (ROS) thus predisposing to oxidative stress disturbances. Many of the clinical and pathophysiological features of IBD, particularly tissue injury (mucosal erosions) and fibrosis have been associated to redox imbalance due to continuous ROS production and a net decrease of antioxidant molecules. Although uncontrolled oxidative stress is destructive in inflammatory conditions, the body's antioxidant defenses can counteract the effects caused by excess of ROS. Antioxidants are protective molecules/compounds toward pro-oxidant molecules. They can be endogenous or/and come from the diet. Endogenous compounds include intracellular enzymatic antioxidants such as superoxide dismutases (SODs), glutathione peroxidase (GPX), and catalase (CAT), intracellular nonenzymatic antioxidant such as glutathione (GSH) and extracellular antioxidants such as vitamins (Vit. A-C-E-B group). GSH is considered the major non-protein low molecular weight defender against oxidative (or redox) stress and the most important cellular thiol buffer. Moreover it acts as cofactor for the antioxidant enzymes GPxs and GST. GSH has been used as a biomarker for inflammation and several studies showed reduced levels of GSH in inflammatory conditions. Experimental colitis models showed decreased GSH levels that can be restored to a normal level by antioxidants supplementation. Also antioxidant enzymes as SODs, CAT and GPxs were found dysregulated in IBD condition. The differences in the regulation of expression of SOD, CAT and GPxs may not only reflect their importance in physiology, but may be also insufficient in removal of ROS under inflammatory conditions such as IBD.

Recently an association between SOD1, CAT and GSHPX1 polymorphisms and the risk of inflammatory bowel disease in the Polish population has been described. Kosaka et al. found a correlation between age of onset and severity of IBD with polymorphisms in SOD2 manganese superoxide dismutase and NAD(P)H quinone oxidoreductase. In this respect, IBD disease can be regarded as multifactorial disease. There are several lines of evidence to suggest that diet is a key player in the onset, perpetuation and management of IBD. The most important evidence linking diet to IBD comes from exclusive enteral nutrition (EEN) that is the primary induction treatment of active paediatric Crohn Disease (CD). Epidemiological evidence associates certain dietary nutrients and components to the increased risk of IBD. There is emerging evidence that some diets, including the Specific Carbohydrate Diet (SCD) and the CD Exclusion Diet (CDED) could treat or prevent subsequent disease flare. Data previously presented induce to the hypothesis that an antioxidant dietetic approach, could have a role in the treatment of IBD. Dietary antioxidants may include ascorbic acid, vitamin E, glutathione, methionine, carotenoids, polyphenolic compounds, selenium and vitamin A. Clinical experience evaluating antioxidant dietetic approach in IBD patients is limited to few studies, mostly investigating the effects of single antioxidants in small number of patients. So far pediatric data regarding the oxidative status in children with IBD have rarely been reported. Collecting data in IBD children and comparing these with adults data, particularly in subjects at diagnosis, would give the unique opportunity to evaluate the role of oxidative stress in IBD pathogenesis. OxIBDiet working hypothesis is that oxidative stress imbalance is a key feature of IBD and the persistence of such imbalance is likely to contribute to the development of complications and more broadly to the evolution of the disease. A comparison between oxidative stress imbalance in children and adults with IBD and controls will address the question whether the stress imbalance is a consequence or a primary event in the inflammatory burden of IBD. Addressing these pathways and targeting the oxidative damage can have potential implications in IBD monitoring and treatment.

This study has been granted by the Italian Ministry of Health (grant RF 2018-12366976)

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of IBD

Exclusion Criteria:

* permanent stoma
* cancer
* cardiovascular disease
* ischemic disease
* Alzheimer's disease
* type 2 diabetes

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2024-06-08 (Actual); Study Completion 2024-12-08 (Estimated)

PRIMARY OUTCOMES:
Blood levels of ROS and glutathione in patients with IBD and controls | Baseline
  Blood levels of ROS will be determined by cytofluorimetry, blood levels of glutathione by spectrofluorimetry
Total antioxidant capacity (Trolox equivalent and ferrous equivalent) in patients with IBD and controls | Baseline
  Trolox equivalent will be assessed by antioxidant assay Kit, ferrous equivalent instead wille require a manual assessment.
Antioxidant enzymes pattern (GST, SOD, GPxs, GR enzyme levels, activity and transcripts) in patients with IBD and controls | Baseline
  Spectrophotometer will be used to assess enzyme levels and activity, cDNA kit to determine enzyme transcripts.
Plasma hydroperoxides and thiobarbituric acid reactive species in patients with IBD and controls | Baseline
  Plasma hydroperoxides will be detected by LPO ELISA kit, thiobarbituric acid reactive species by TBARS assay kit.
Urine oxidized guanines (8-OHdG, 8-OHG e guanosine) levels in patients with IBD and controls | Baseline
  DNA/RNA oxydate damage kit will be used to study urine oxidized guanines levels.

SECONDARY OUTCOMES:
Polymorphisms of genes implicated in oxidative stress defense (SOD1, SOD2, SOD3; GPX1, GPX2, GPX3; GPX4; GPX5; GSTA1; GSTA2; GSTM1; GSTM2; GSTM3; GSTP1; GSTO1; NQ01 NQ02; NOX1; NOX3; NOX4 and NOX5 genes) in patients with IBD and controls | Baseline
  Genetic polymorphisms will be studied by next generation sequencing

OTHER OUTCOMES:
Blood levels of ROS and glutathione in patients with IBD after a specific antioxidant dietary treatment | 12 weeks
  Blood levels of ROS will be determined by cytofluorimetry, blood levels of glutathione by spectrofluorimetry at baseline and after 12 weeks of dietary treatment.
Total antioxidant capacity (Trolox equivalent and ferrous equivalent) in patients with IBD after a specific antioxidant dietary treatment | 12 weeks
  Trolox equivalent will be assessed by antioxidant assay Kit, ferrous equivalent instead wille require a manual assessment at baseline and after 12 weeks of dietary treatment.
Antioxidant enzymes pattern (GST, SOD, GPxs, GR enzyme levels, activity and transcripts) in patients with IBD after a specific antioxidant dietary treatment | 12 weeks
  Spectrophotometer will be used to assess enzyme levels and activity, cDNA kit to determine enzyme transcripts at baseline and after 12 weeks of dietary treatment
Plasma hydroperoxides and thiobarbituric acid reactive species in patients with IBD after a specific antioxidant dietary treatment | 12 weeks
  Plasma hydroperoxides will be detected by LPO ELISA kit, thiobarbituric acid reactive species by TBARS assay kit at baseline and after 12 weeks of dietary treatment.
Urine oxidized guanines (8-OHdG, 8-OHG e guanosine) levels in patients with IBD after a specific antioxidant dietary treatment | 12 weeks
  DNA/RNA oxydate damage kit will be used to study urine oxidized guanines levels at baseline and after 12 weeks of dietary treatment
PUCAI in pediatric patients with RCU after a specific antioxidant dietary treatment | 12 weeks
  PUCAI score will be recorded at baseline and after 12 weeks of dietary treatment
PCDAI in pediatric patients with CD after a specific antioxidant dietary treatment | 12 weeks
  PCDAI score will be recorded at baseline and after 12 weeks of dietary treatment
Phisician Global Assessment (PGA) score in patients with IBD after a specific antioxidant dietary treatment | 12 weeks
  PGA score will be recorded at baseline and after 12 weeks of dietary treatment
Calprotectin levels in patients with IBD after a specific antioxidant dietary treatment | 12 weeks
  Calprotectin levels will be analyzed in stool samples collected at baseline and after 12 weeks of dietary treatment
Harvey-Bradshaw score in adult patients with CD after a specific antioxidant dietary treatment | 12 weeks
  Harvey-Bradshaw score will be recorded at baseline and after 12 weeks of dietary treatment
Mayo score in adult patients with RCU after a specific antioxidant dietary treatment | 12 weeks
  Mayo score will be recorded at baseline and after 12 weeks of dietary treatment
PedQoL score in pediatric patients with IBD after a specific antioxidant dietary treatment | 12 weeks
  PedQoL score will be recorded at baseline and after 12 weeks of dietary treatment
QoL score in adult patients with IBD after a specific antioxidant dietary treatment | 12 weeks
  QoL score will be recorded at baseline and after 12 weeks of dietary treatment

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Catassi, Professor, Principal Investigator — Università Politecnica delle Marche
Locations (2):
- Italy (2):
  - SOD Clinica Pediatrica, Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona
  - SOD Clinica di Gastroenterologia, Epatologia ed Endoscopia Digestiva, Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after deidentification will be shared
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata.

REFERENCES:
- [Background] Kolho KL, Ainamo A. Progress in the treatment and outcome of pediatric inflammatory bowel disease patients. Expert Rev Clin Immunol. 2016 Dec;12(12):1337-1345. doi: 10.1080/1744666X.2016.1201422. Epub 2016 Jun 29. PMID 27322874
- [Background] Sigall-Boneh R, Levine A, Lomer M, Wierdsma N, Allan P, Fiorino G, Gatti S, Jonkers D, Kierkus J, Katsanos KH, Melgar S, Yuksel ES, Whelan K, Wine E, Gerasimidis K. Research Gaps in Diet and Nutrition in Inflammatory Bowel Disease. A Topical Review by D-ECCO Working Group [Dietitians of ECCO]. J Crohns Colitis. 2017 Dec 4;11(12):1407-1419. doi: 10.1093/ecco-jcc/jjx109. PMID 28961811
- [Background] Gatti S, Galeazzi T, Franceschini E, Annibali R, Albano V, Verma AK, De Angelis M, Lionetti ME, Catassi C. Effects of the Exclusive Enteral Nutrition on the Microbiota Profile of Patients with Crohn's Disease: A Systematic Review. Nutrients. 2017 Aug 4;9(8):832. doi: 10.3390/nu9080832. PMID 28777338
- [Result] Tian T, Wang Z, Zhang J. Pathomechanisms of Oxidative Stress in Inflammatory Bowel Disease and Potential Antioxidant Therapies. Oxid Med Cell Longev. 2017;2017:4535194. doi: 10.1155/2017/4535194. Epub 2017 Jun 28. PMID 28744337
- [Result] Pereira C, Gracio D, Teixeira JP, Magro F. Oxidative Stress and DNA Damage: Implications in Inflammatory Bowel Disease. Inflamm Bowel Dis. 2015 Oct;21(10):2403-17. doi: 10.1097/MIB.0000000000000506. PMID 26193347
- [Result] Mrowicka M, Mrowicki J, Mik M, Wojtczak R, Dziki L, Dziki A, Majsterek I. Association between SOD1, CAT, GSHPX1 polymorphisms and the risk of inflammatory bowel disease in the Polish population. Oncotarget. 2017 Nov 27;8(65):109332-109339. doi: 10.18632/oncotarget.22675. eCollection 2017 Dec 12. PMID 29312611
- [Result] Kosaka T, Yoshino J, Inui K, Wakabayashi T, Kobayashi T, Watanabe S, Hayashi S, Hirokawa Y, Shiraishi T, Yamamoto T, Tsuji M, Katoh T, Watanabe M. Involvement of NAD(P)H:quinone oxidoreductase 1 and superoxide dismutase polymorphisms in ulcerative colitis. DNA Cell Biol. 2009 Dec;28(12):625-31. doi: 10.1089/dna.2009.0877. PMID 19715479
- [Result] Dryden GW, Lam A, Beatty K, Qazzaz HH, McClain CJ. A pilot study to evaluate the safety and efficacy of an oral dose of (-)-epigallocatechin-3-gallate-rich polyphenon E in patients with mild to moderate ulcerative colitis. Inflamm Bowel Dis. 2013 Aug;19(9):1904-12. doi: 10.1097/MIB.0b013e31828f5198. PMID 23846486
- [Result] Kolacek M, Muchova J, Dvorakova M, Paduchova Z, Zitnanova I, Cierna I, Orszaghova Z, Szekyova D, Jajcaiova-Zednickova N, Kovacs L, Durackova Z. Effect of natural polyphenols (Pycnogenol) on oxidative stress markers in children suffering from Crohn's disease--a pilot study. Free Radic Res. 2013 Aug;47(8):624-34. doi: 10.3109/10715762.2013.807508. Epub 2013 Jun 13. PMID 23710677
- [Result] Rastegarpanah M, Malekzadeh R, Vahedi H, Mohammadi M, Elahi E, Chaharmahali M, Safarnavadeh T, Abdollahi M. A randomized, double blinded, placebo-controlled clinical trial of silymarin in ulcerative colitis. Chin J Integr Med. 2015 Dec;21(12):902-6. doi: 10.1007/s11655-012-1026-x. Epub 2012 Apr 11. PMID 22528757
- [Result] Aghdassi E, Wendland BE, Steinhart AH, Wolman SL, Jeejeebhoy K, Allard JP. Antioxidant vitamin supplementation in Crohn's disease decreases oxidative stress. a randomized controlled trial. Am J Gastroenterol. 2003 Feb;98(2):348-53. doi: 10.1111/j.1572-0241.2003.07226.x. PMID 12591053